CLINICAL TRIAL: NCT01529060
Title: A Double-Blind, Randomized, Placebo-Controlled, Crossover Trial of Phenylbutyrate in the Treatment of Maple Syrup Urine Disease
Brief Title: Phenylbutyrate Therapy for Maple Syrup Urine Disease
Acronym: MSUD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brendan Lee (Other)
Responsible Party: Sponsor-Investigator, Brendan Lee, Professor, Molecular and Human Genetics, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H-28463
Record Dates: First submitted 2012-02-06; First posted 2012-02-08 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Maple Syrup Urine Disease
Keywords: phenylbutyrate; MSUD; Buphenyl-TM
MeSH Terms: conditions — Maple Syrup Urine Disease | interventions — Phenylbutyrates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phenylbutyrate (Active Comparator): Study Drug
  Interventions: Drug: Phenylbutyrate
- Inactive Powder (Placebo Comparator): Placebo powder
  Interventions: Drug: Placebo powder

INTERVENTIONS:
Drug: Phenylbutyrate — Dosage of phenylbutyrate powder will be 500 mg/kg/day in patients weighing less than 20kg and 10 g/m2/day in larger patients in four divided doses per day, the standard UCD dose studied in our preliminary studies, for 14 days.
  Other Names: Buphenyl-TM
  Arms: Phenylbutyrate
Drug: Placebo powder — Dosage of inactive placebo powder will be 500 mg/kg/day in patients weighing less than 20kg and 10 g/m2/day in larger patients in four divided doses per day for 14 days. Subjects will receive the same amount of powder for each arm of the study.
  Arms: Inactive Powder

SUMMARY:
The investigators have learned in past research that the drug phenylbutyrate can decrease the amounts of branched chain amino acids and their byproducts in the bloodstreams of healthy volunteer patients and also patients with certain disorders of protein breakdown including maple syrup urine disease. Through this study, the investigators will try to find out how well phenylbutyrate (NaPBA), also known by name brand "Buphenyl-TM", decreases BCAA and branched chain keto chain acids in the blood of patients with MSUD. The investigators hope is that through this research the investigators will be better able to treat these patients.

Subjects with MSUD will take phenylbutyrate (NaPBA) in powder form for a two-week treatment period and powder placebo, a substance with no effect on the body, for a two-week treatment period. They will be given the same amount of powder and undergo the same laboratory testing during both of the two-week treatment periods. The results will be compared once the study is over.

DETAILED DESCRIPTION:
Maple syrup urine disease is a severe inborn error of amino acid metabolism caused by deficiency of the mitochondrial branched-chain alpha-ketoacid dehydrogenase complex (BCKDC) resulting in the accumulation of branched-chain amino acids (BCAA) (isoleucine, leucine, and valine) and their corresponding branched-chain alpha-ketoacids (BCKA) [alpha-keto-beta-methylvalerate (KMV), alpha-ketoisocaproate (KIC), and alpha-ketoisovalerate(KIV)] in tissues and plasma. The disorder typically manifests with potentially lethal episodes of intoxication presenting with acute neurological deterioration, feeding problems, weight loss, and a maple syrup odor to the urine. Current treatment is based on dietary manipulations with protein restriction and a synthetic formula with reduced BCAA content. However, mental and social impairment are still present in the majority of these patients in spite of dietary management.

Our study seeks to investigate the potential small molecule inhibition of the kinase that regulates BCKDC by applying a novel activity of sodium phenylbutyrate (NaPBA), in MSUD. Sodium phenylbutyrate is has been used to treat patients with urea cycle disorders (UCDs). In our extensive studies with UCDs, we noted that patients on therapy with NaPBA had decreased plasma levels of BCAA. This led us to hypothesize that NaPBA has effects on BCAA metabolism.

This will be a single-site, randomized, active-controlled, double-blind, cross-over study designed to enroll subjects with MSUD. Subjects will be randomly assigned to receive either sodium phenylbutyrate (PB) or placebo for 2 weeks, and then crossed over to receive the other treatment for 2 weeks.

If study findings show sodium phenylbutyrate lowers BCAA and BCKA levels in these patients, it may prove to be an effective adjunct treatment for these patients. A treatment option that could prevent or decrease the accumulation of BCAA and BCKA during states of catabolism induced by fasting or intercurrent illnesses, and thereby minimize or prevent the neurologic sequelae and loss of human potential that result, would greatly benefit society.

ELIGIBILITY:
Inclusion Criteria:

* Must be 3 years or older at enrollment.
* Must have a diagnosis of maple syrup urine disease (MSUD) confirmed by the presence of plasma alloisoleucine (>5 micromol/L) and/or genetic testing showing mutations in both alleles of any subunit of BCKDHA (E1alpha subunit gene, MSUD type 1A), BCKDHB (E1beta subunit gene, MSUD type 1B), or DBT (E2 subunit gene, MSUD type 2).
* Participants must have a history of compliance to diet and treatment.
* Signed informed consent by subject and/or subject's legally acceptable representative.
* Must be capable of completing study procedures, including taking oral or G- tube medication.
* Negative pregnancy test for all females of childbearing potential.
* All females of childbearing potential and all sexually active males must agree to use an acceptable method of contraception throughout the study. Appropriate contraceptive methods include hormonal contraceptives (oral, injected, implanted, or transdermal), tubal ligation, intrauterine device, hysterectomy, vasectomy, or double barrier methods. Abstinence is an acceptable form of birth control, though appropriate contraception must be used if the subject becomes sexually active.

Exclusion Criteria:

* May not have used sodium phenylbutyrate within 30 days of Visit 1.
* May not have an active infection (viral or bacterial) or any condition which may exacerbate their MSUD causing metabolic decompensation.
* Cannot have any clinical or laboratory abnormality of Grade 3 or greater according to the Common Terminology Criteria for Adverse Events v3.0 (CTCAE) (or for conditions not covered by the CTCAE, a severe or life-threatening toxicity).
* May not have taken any medications known to significantly affect renal clearance or to increase protein catabolism within the 24 hours prior to Visit 1.
* May not participate if they have a known hypersensitivity to phenylacetate or phenylbutyrate or creatinine levels 1.5 times or more ULN.
* Since a total of 53 mL will be drawn over Days 14 and 15 of both treatment periods, only subjects weighing more than 30 pounds can be enrolled.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2017-09-02 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Lee, M.D., Ph.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- See also: Baylor College of Medicine Website — http://www.bcm.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Phenylbutyrate First and Placebo Second Group: Individuals randomized to this group received phenylbutyrate powder (500 mg/kg/day in patients weighing less than 20kg and 10 g/m2/day in larger patients in 3 divided doses per day) for 14 days (week 1 and week 2) and then crossed over to receive placebo powder in identical doses for the next 14 days (Week 3 and week 4)
- Placebo First and Phenylbutyrate Second Group: Individuals randomized to this group received first received placebo powder for 14 days (week 1 and week 2) and then were crossed over to receive phenylbutyrate (500 mg/kg/day in patients weighing less than 20kg and 10 g/m2/day in larger patients in 3 divided doses per day) for 14 days (week 3 and week 4) week 4).
Period: Overall Study
Arm/Group | Phenylbutyrate First and Placebo Second Group | Placebo First and Phenylbutyrate Second Group
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Anaysis population is same as the the one depicted in Participant Flow
Groups:
- Phenylbutyrate First and Placebo Second: Individuals randomized to this group received phenylbutyrate (500 mg/kg/day in patients weighing less than 20kg and 10 g/m2/day in larger patients in divided doses per day) for 14 days (week 1 and week 2) and then crossed over to receive placebo powder in identical doses for the next 14 days (Week 3 and week 4)
- Placebo First and Phenylbutyrate Second: Individuals randomized to this group received first received placebo powder for 14 days (week 1 and week 2) and then were crossed over to receive phenylbutyrate (500 mg/kg/day in patients weighing less than 20kg and 10 g/m2/day in larger patients in 3 divided doses per day) for 14 days (week 3 and week 4) week 4).
- Total: Total of all reporting groups
Arm/Group | Phenylbutyrate First and Placebo Second | Placebo First and Phenylbutyrate Second | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Full Range); unit: years] | 23 [15 to 43] | 23 [10 to 45] | 23 [10 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 3 | 6 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic Categories: Not Hispanic or Latino | 8 | 9 | 17
  Ethnic Categories: Hispanic or Latino | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19
  Canada | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: 0-24 Hour AUC Leucine (Samples Collected at 0, 2, 4, 8, 12, 16, 20, and 24 Hours)
Description: Total Leucine exposure over 24 hours was calculated by serial blood draws at times 0, 2, 4, 8, 12, 16, 20, and 24 hours
Time Frame: 24 Hours
Measure: Mean (Standard Deviation); unit: micromoles*hour/L
Groups:
- Phenylbutyrate: Cumulative results when individuals were treated with phenylbutyrate
- Placebo First and Phenylbutyrate Second Group: Cumulative results from when individuals were treated with placebo
Arm/Group | Phenylbutyrate | Placebo First and Phenylbutyrate Second Group
Number analyzed (Participants) | 20 | 20
micromoles*hour/L | 6217 (5168) | 4616 (4106)

2. Primary Outcome: Leucine CMax 0-24 Hours
Description: Maximal leucine concentration in 0-24 hours
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Micromoles/L
Groups:
- Placebo: Cumulative results when individuals were treated with placebo
Arm/Group | Phenylbutyrate | Placebo
Number analyzed (Participants) | 20 | 20
Micromoles/L | 361 (244) | 295 (211)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 14 days of Treatment period 1 and 14 days of treatment period 2
Arm/Group | Phenylbutyrate | Inactive Powder
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 19/20 | 16/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phenylbutyrate (N=20) | Inactive Powder (N=20)
Oral or Nasal Complaints (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 4 (4)
Labs (Blood and lymphatic system disorders) | 19 (19) | 16 (16)
Gastrointestinal Symptoms (Gastrointestinal disorders) | 16 (16) | 7 (7)
Neurological Complaints (Nervous system disorders) | 7 (7) | 7 (7)
Muscular Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Minor Skin Complaints (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Urine Odor (Renal and urinary disorders) | 1 (1) | 1 (1)
Menstral Cramps (Reproductive system and breast disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT01529060/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT01529060/SAP_001.pdf